CLINICAL TRIAL: NCT03396783
Title: Characterization of the Immunological Profile Patients With Post-polio Syndrome in Comparison With These Control Subjects
Brief Title: Characterization of the Immunological Profile Patients With Post-polio Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: RECHMPL16_0080; UF9753 (Other: UH Montpellier)
Record Dates: First submitted 2017-11-09; First posted 2018-01-11 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis Sequelae
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPP (Experimental): during the visit, nurse will make a blood test for biological and immunological analysis, electromyogram and walk test
  Interventions: Biological: blood test; Other: electromyogram and walk test
- Control (Other): during the visit, nurse will make a blood test for biological and immunological analysis
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — during the visit, nurse will make a blood test for biological and immunological analysis
Other: electromyogram and walk test — during the visit, measuring the amount of functional motor units at the muscular level and the distance traveled during a 2 minute walk
  Arms: SPP

SUMMARY:
Many patients with polio sequelae have persistent and progressive worsening more than 15 years after the initial damage, with loss of muscle strength, asthenia and musculoskeletal pain. In these patients, there is a denervation process associated with insufficient reinnervation. The frequency of this syndrome post-polio (SPP) is of the order of 20 to 60% according to the studies. In the literature, several studies have advanced the hypothesis of immune dysregulation to this late degradation, with greater expression of pro-inflammatory cytokines, and abnormal phenotypic expression of T cells in the bloodstream. In this context, the use of immunomodulatory immunoglobulin IV treatment was studied several times, with no significant result on pain, fatigue and muscle strength scores. In the absence of significant efficacy of immunoglobulin treatment, the objective of this study is therefore to define the immunological profile of patients with post-polio syndrome, compared with control subjects, in order to support the pathophysiology of this syndrome. to study the possible presence of an inflammatory syndrome associated with this syndrome. On the other hand, depending on the results found, referral to targeted therapies could be considered.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Post-polio Syndrome :

* age ≥ 18 years
* meeting the definition of the SPP according to the criteria of Halstead et al. (1995)

Controlled subjects :

* age ≥ 18 years
* matched on sex and age (+/- 5 years) with subjects with PPS

Exclusion Criteria:

* intercurrent neurological pathology,
* uncontrolled cardiovascular risk factors
* pulmonary comorbidity
* endocrine disorders
* systemic inflammatory pathology, autoimmune disease, dry syndrome,
* renal failure
* anti-inflammatory treatment in progress or in the previous month, or immunoregulatory aim whatever its nature,
* patients with SPP who received polyvalent IV immunoglobulins in the 3 years prior to inclusion, or taking anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
cytokines blood concentrations | blood sample during inclusion visit
lymphocytes blood concentrations | blood sample during inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAFFONT, Principal Investigator — UH Montpellier
Locations (1):
- CHRU Lapeyronie, Montpellier, Herault, France